CLINICAL TRIAL: NCT04709471
Title: Electronic Nicotine Delivery Systems' Influence on Combustible Cigarette Smoking and Demand: A Randomized Controlled Trial
Brief Title: E-cigarette Nicotine Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Elias Klemperer, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001093
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-05

CONDITIONS: Nicotine Dependence; Electronic Cigarette Use; Cigarette Smoking
Keywords: Cigarettes; Electronic nicotine delivery systems; Electronic cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Cigarette Smoking | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Switch to low nicotine e-cigarettes (Experimental): Switch to e-cigarettes containing 60% of baseline e-cigarette nicotine content.
  Interventions: Drug: Nicotine; Device: Juul e-cigarette
- Reduce number of e-cigarette pods (Experimental): Reduce e-cigarette use to 60% of baseline number of pods per week.
  Interventions: Drug: Nicotine; Behavioral: Reduction
- Use e-cigarettes as usual (No Intervention): Continue using usual nicotine e-cigarettes as usual.

INTERVENTIONS:
Drug: Nicotine — Participants will reduce their nicotine intake
  Arms: Reduce number of e-cigarette pods; Switch to low nicotine e-cigarettes
Device: Juul e-cigarette — Participants will switch to Juul pods containing less nicotine
  Arms: Switch to low nicotine e-cigarettes
Behavioral: Reduction — Participants will reduce the number of Juul pods that they use
  Arms: Reduce number of e-cigarette pods

SUMMARY:
This is a pilot randomized controlled trial (RCT) with the overarching aim of testing the influence of reducing electronic nicotine delivery system (ENDS) use or nicotine on addiction and combustible cigarette (CC) smoking among dual users. Specifically, the investigators will conduct a 4-week pilot RCT in which dual users who are not motivated to quit either product in the near future are randomized to A) abruptly switch to low nicotine ENDS pods, B) abruptly reduce number of usual nicotine ENDS pods, or C) use ENDS as usual (control). The investigators adapted a protocol used in a prior study to assign participants to switch to ENDS pods with less nicotine or reduce number of ENDS pods in this trial. Specifically, the investigators will provide all participants with ENDS pods during the study period and instruct them to only use ENDS provided by the study. Participants in reduced nicotine condition will switch from usual nicotine (5% JUUL) to low nicotine ENDS (3% nicotine JUUL) pods. Participants in the reduced use condition will continue to use usual nicotine ENDS (5% nicotine JUUL) pods but reduce use to 60% of their baseline number of pods per week. Participants in the control condition will use usual nicotine ENDS (5% nicotine JUUL) pods as usual.

DETAILED DESCRIPTION:
Background Use of Electronic Nicotine Delivery Systems (ENDS) has increased substantially in the past decade, and nearly 70% of ENDS users also smoke cigarettes (i.e., dual users). There is evidence that ENDS can be used as an effective smoking cessation aid. However, most dual users use ENDS intermittently, which does not appear to promote smoking cessation. ENDS use appears to be associated with increased overall nicotine addiction in some dual users and could perpetuate or increase combustible cigarette (CC) smoking. These concerns have contributed to policy changes to restrict ENDS use. For example the FDA's Center for Tobacco Products finalized a rule to regulate ENDS and could reduce the amount of nicotine in ENDS. Further, some states have begun to restrict access to ENDS. Market restrictions, FDA warning labels, and public education messaging have the potential to reduce ENDS consumption. Little is known, however, regarding the mechanisms of change in ENDS use that could affect nicotine addiction and CC smoking in dual users. Thus, the investigators are conducting a pilot randomized controlled trial (RCT) to test how change in ENDS nicotine (i.e. pharmacology) and change in frequency of ENDS use (i.e., behavior) affects nicotine addiction and CC smoking among dual users. Findings will inform understanding of how change in ENDS use contributes to nicotine addiction and how regulation that results in reduced nicotine consumption from ENDS could affect tobacco use among dual users.

Both pharmacological and behavioral factors contribute to nicotine dependence and thus could be mechanisms by which change in ENDS affects addiction among dual users. Prior research identified that switching to low nicotine CCs (i.e., change in pharmacology) and reduction in number of CCs (i.e., change in behavior) independently reduced nicotine dependence and demand for cigarettes within-participants over time. Similarly, observational data indicate that self-selected use of lower nicotine content ENDS (i.e., pharmacology) and less frequent vaping (i.e., behavior) appear to be associated with lower overall nicotine dependence among dual users. However, there is a lack of experimental research on whether change in ENDS nicotine content or frequency of use affects overall nicotine dependence among dual users.

Specific Aims

Primary Aim 1: To assess the feasibility of abruptly switching to low nicotine ENDS pods or abruptly reducing number of ENDS pods.

Aim 2: To assess the influence of switching to reduced nicotine ENDS compared to ENDS use as usual on CC smoking and nicotine dependence.

Aim 3: To assess the influence of reducing number of usual nicotine ENDS pods compared to ENDS use as usual on CC smoking and nicotine dependence.

Secondary Aim 4: To assess the influence of switching to reduced nicotine ENDS pods compared to reducing number of usual nicotine ENDS pods on CC smoking and nicotine dependence.

Methodology The procedures are based on a methodology demonstrated to be feasible in a prior research. Potential participants who screen eligible will complete a videoconference call with study personnel to 1) display their photo ID to confirm their identity, 2) display their Juul device to confirm that they use Juul products, and 3) review the consent form. Participants will provide written consent using the REDCap e-consent procedure. Consenting participants will answer brief nightly questionnaires about the amount they smoke CCs and use JUUL during a baseline week (week 0). During the baseline week (week 0) research personnel will mail participants a personal iCO Smokerlyzer (https://www.covita.net/ico-overview/) for remote breath carbon monoxide (CO) measurement. Research personnel will also mail a pregnancy test to all female participants of reproductive potential (see Inclusion/Exclusion criteria section below). At the end of the baseline week (week 0), participants will be emailed a link to a REDCap survey to answer demographic and tobacco-related baseline questionnaires, to report their breath CO level using their personal iCO Smokerlyzer, and, for women of reproductive potential, to report the results of their pregnancy test. Women who are pregnant or plan to become pregnant will not be eligible to participate in this study and will be removed from this study if they become pregnant. At the end of the baseline (week 0) REDCap survey, participants will be randomly assigned to A) abruptly switch to low nicotine ENDS pods, B) abruptly reduce number of usual nicotine ENDS pods per week, or C) use ENDS as usual. After completing the baseline REDCap survey, participants will be mailed their study JUUL pods according to their condition. All participants will continue to complete brief nightly questionnaires throughout the remaining 4-week study period. In addition, participants will provide breath CO samples remotely using a personal iCO Smokerlyzer provided by the study and complete tobacco related questionnaires remotely via REDCap at the end of each week throughout the study period.

Participants will use their own JUUL products during baseline (week 0) and will be instructed to only use JUUL products provided by the study throughout weeks 1 through 4. In order to increase the validity of participants' self-reported adherence to study ENDS products (i.e., feasibility), the investigators will inform participants that self-reported noncompliance will not influence their payment or future participation. At the end of week 0, the investigators will provide participants with 4-week supplies of JUUL pods based on their assigned condition and the number of pods they used during baseline (i.e. week 0) via mail. The investigators will provide participants who are randomized to switch to low nicotine ENDS with 100% of the number of JUUL pods/week used during the baseline week, but all JUUL pods provided will have a nicotine content reduced to 60% of baseline (i.e., 3% nicotine JUUL pods). The investigators will provide participants who are randomized to reduce number of ENDS with approximately 60% of the number of JUUL pods/week used during the baseline week, and all JUUL pods provided will have the regular nicotine content (i.e., 5% nicotine JUUL pods). The investigators chose to reduce participants' number of JUUL pods to approximately 60% of baseline to match the 60% reduction in nicotine in the group assigned to switch from usual (5%) to low (3%) nicotine JUUL pods. In addition, a similar magnitude of cigarette reduction was feasible in a prior trial. Finally, participants randomized to use ENDS as usual (control condition) will be provided with 100% of their baseline number of JUUL pods/week containing regular nicotine content (5%). Participants in all conditions will have the option to choose their preferred flavor of JUUL pods among the flavors sold legally in Vermont when they are participating. The investigators will clearly and explicitly state that they are not requiring participants to change CC smoking. Given the potential for compensatory CC smoking during the study period, the study will have a data and safety monitoring board (DSMB) review the study procedures and monitor participants' safety as necessary.

At the end of week 4 the investigators will provide all participants with advice to quit all tobacco products. They will also provide all participants a referral to the national quitline for information on the benefits of quitting tobacco. In addition they will offer to mail a one-month supply of nicotine replacement therapy (NRT) to participants who confirm they have no contraindications for NRT to help them quit. Thus participants interested in NRT will complete a brief screener via REDCap at the end of week 4. Participants who endorse a) Recent heart attack (in last month), b) Heart disease that is untreated, c) Arrhythmia or irregular heartbeat, d) High blood pressure not controlled by medications, e) An allergy to adhesive tape, f) Skin problems that require treatment, or g) Stomach ulcer or diabetes will receive a referral to the quitline but will not be eligible for NRT. The investigators will not provide any participants with ENDS products after week 4 of the study period. Finally, all participants will complete a web-based follow-up survey and provide a breath CO sample 4 weeks after study completion (i.e., 8 weeks after randomization) to assess tobacco use, ENDS use, quit attempts, and behavioral economic measures.

ELIGIBILITY:
Eligibility criteria include at least 21 years old, use e-cigarettes and tobacco cigarettes regularly, not planning to quit in the near future, and not pregnant, breastfeeding or planning to become pregnant or breastfeed in the next 2 months.

Additional criteria will be evaluated to assess for eligibility.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | Baseline and the four week reduction period
  The investigators will assess compliance with study e-cigarettes and compare the percent non-study e-cigarette use between conditions to determine which behavior-changing strategy is more feasible.
Combustible cigarette smoking | Baseline and the four week reduction period
  The investigators will compare change in number of cigarettes per day between conditions.
Cigarette dependence | Baseline and the four week reduction period
  The investigators will compare change in cigarette dependence between conditions using the PATH dependence measure.
E-cigarette dependence | Baseline and the four week reduction period
  The investigators will compare change in e-cigarette dependence between conditions using the PATH dependence measure.

SECONDARY OUTCOMES:
Cigarette demand | Baseline and the four week reduction period
  The investigators will compare change in cigarette demand using the the Brief Assessment of Cigarette Demand task.
E-cigarette demand | Baseline and the four week reduction period
  The investigators will compare change in e-cigarette demand using a version of the the Brief Assessment of Cigarette Demand task adapted for e-cigarettes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No